CLINICAL TRIAL: NCT05459948
Title: Medacta GMK® SpheriKA and Kinematic Alignment Technique Multicenter, Post-Market Outcome Study
Brief Title: The Medacta GMK SpheriKA Post-Marketing Surveillance Study
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P.02.025.02
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-03

CONDITIONS: Arthropathy; Knee Replacement
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Device: GMK SpheriKA — The first objective is to study the FJS of patients who were implanted a "GMK® SpheriKA" knee prosthesis using the kinematic alignment technique

SUMMARY:
This is a Post-Marketing Surveillance of GMK SpheriKA knee stem prosthesis.

DETAILED DESCRIPTION:
The aim of the current study is to collect clinical and radiological data to monitor the performances of the "GMK® SpheriKA" Knee Prosthesis implanted via the kinematic alignment technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign the informed consent.
* Patients able to comply with follow-up requirements, including postoperative weight-bearing restrictions and self-evaluations.
* Patients 18 - 80 years of age at the time of surgery.
* Patients requiring a primary total knee replacement (on label use).
* Patients with intact collateral ligaments.

Exclusion Criteria:

* Patients with inflammatory arthritis.
* Morbidly obese patients, with a body mass index (BMI) > 40.
* Patients with a history of total or unicompartmental reconstruction of the affected joint.
* Patients that have had a high tibial osteotomy or femoral osteotomy.
* Patients with neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
* Patients with a systemic or metabolic disorder leading to progressive bone deterioration.
* Patients that are immunologically compromised or receiving chronic steroids (> 30 days).
* Patients whose bone stock is compromised due to disease or infection, unable to provide adequate support and/or fixation to the prosthesis.
* Patients with an active or suspected latent infection in or surrounding the knee joint.
* Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 281 participants are planned for the entire project (all sites combined). Patients requiring "GMK® SpheriKA" implanted via the kinematic alignment technique will be informed and enrolled during the preoperative visit.
  The study is conducted as standard of care treatment and participants will receive the same treatment and undergo the same postoperative assessments as non-participants.
Sampling Method: Probability Sample
Enrollment: 281 (Estimated)
Dates: Start 2022-07-30 (Actual); Primary Completion 2035-05 (Estimated); Study Completion 2035-05 (Estimated)

PRIMARY OUTCOMES:
Primary objective will be evaluated with the Forgotten Joint score (FJS). | 6 weeks, from 1 to 10 years annually
  study the efficacy of the treatment to make the patient forget the presence of the artificial joint in everyday life.
  The Forgotten Joint Score assessment consists of 12 questions and is scored on a 0-100 scale. The higher the score, the less the patient is aware of their affected joint when performing daily activities

SECONDARY OUTCOMES:
patient-reported outcomes 1 | 6 weeks, from 1 to 10 years annually
  Oxford Knee Score: The OKS is a patient reported outcome measure that consists of 12 questions about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks
Satisfaction and Expectations questionaires | 6 weeks, from 1 to 10 years annually
  Satisfaction and Expectations questionaires
  Patient reported satisfaction and expectations answering some questions of the "satisfaction and expectation knee society score", the goal is to collect all final answers and have an overview on how the patient feels.
  "Patient Expectations" is a three-question fifteen-point scale that is collected pre-operatively and post-operatively.
  "Patient Satisfaction" is a five-question 40-point scale that is collected preoperatively and at each follow-up visit.
Radiological outcomes | pre-op, 6weeks, 1, 2,5,10 years
  Radiological assessment including implant positioning, presence of radiolucent lines, subsidence, migration of components, presence of heterotopic ossifications or osteolysis
Adverse events | during surgical operation, 6weeks, 1,2,5,10 years
  Adverse events (type of complications, dependent or not from the device etc)
Limb alignment | on preoperative and 6-week x-rays
  Limb alignment will be measured: mMPTA (°), mLDFA (°) and joint line (HKA) will be recorded.
  HKA = Hip-Knee-ankle angle measured in degrees mMPTA = mechanical medial proximal tibial angle measured in degrees mLDFA = mechanical lateral distal femoral angle measured in degrees
Lateral uncoverage of the anterior femoral resection | During Surgical Operation
  Measurement of the lateral uncoverage of the anterior femoral resection measured in mm

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - Centre de l'Arthrose, Mérignac
  - Clinique de l'Union, Saint-Jean
- Humanitas Castelli, Bergamo, Italy
- Gelenkzentrum Winterthur, Winterthur, Switzerland